CLINICAL TRIAL: NCT01849614
Title: Prospective Pilot Study of Assessment of Breath Hold as a Means to Mitigate the Risk of Radiation-associated Reductions in Regional Cardiac Perfusion in Patients With Left-sided Breast Cancer
Brief Title: Assessment of Ability of Breath Hold for Left-sided Breast Cancer Radiation Therapy to Reduce Side Effects to Heart
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1239
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient group: Women with left-sided breast cancer
  Interventions: Other: Cardiac SPECT perfusion scan

INTERVENTIONS:
Other: Cardiac SPECT perfusion scan — A SPECT cardiac perfusion scan provides a three-dimensional map of blood flow to the heart tissue. The scan will be taken at rest only.

SUMMARY:
The purpose of this research study is to demonstrate that Deep Inspiration Breath Hold (DIBH), the technique used at the University of North Carolina (UNC) for left-side breast cancer radiation therapy, can reduce side effects to the heart.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate the rate of radiation-associated regional myocardial perfusion defects in patients 6 months after breast/chestwall radiation with DIBH for left-sided breast cancer. Cardiac perfusion will be assessed using SPECT cardiac perfusion scans pre- and 6 months post-radiation.

ELIGIBILITY:
Inclusion Criteria:

* signed an Institutional Review Board (IRB)-approved informed consent document for protocol
* age >= 18 years
* histologically confirmed left-sided breast cancer scheduled to undergo curative intent radiation treatment post lumpectomy or mastectomy
* stage 0-III left-sided breast cancer (including DCIS)
* SPECT score of 0 at baseline
* radiation oncologist agrees target volume coverage will not be compromised via use of the DIBH technique along with conformal field shaping

Exclusion Criteria:

* active cardiac disease, defined as a history of angina, arrhythmias, myocardial infarction, congestive heart failure, or any other cardiac condition, which in the opinion of the treating physician would make this protocol unreasonably hazardous for the patient
* symptomatic pulmonary disease currently requiring regular medication including but not restricted to bronchodilators
* concurrent chemotherapy
* prior receipt of mediastinal radiation therapy
* pregnant or lactating women
* inability to understand and follow breathing instructions for the DIBH procedure

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with left-sided breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac perfusion | 6-months post radiation
  Cardiac perfusion will be assessed using SPECT cardiac perfusion scans pre- and 6 months post-radiation. Any post-radiation summed-rest score (SRS) > 0 will be counted as a perfusion defect in the calculation of the perfusion defect rate.

SECONDARY OUTCOMES:
Wall-motion abnormalities | 6-months post-treatment
  The incidence of wall-motion abnormalities will be assessed using SPECT in the same 12 segment scoring system used to quantify perfusion. Wall-motion abnormalities will be recorded as present or absent in each cardiac segment. When present, wall-motion abnormalities wil be classified as gypokinetic, akinetic, or dyskinetic. The extent of wall involvement (small or large portion) will be described as mild or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Zagar, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States